CLINICAL TRIAL: NCT01362439
Title: Efficacy and Tolerability of Flexible Doses of Paliperidone ER in Symptomatic Subjects With Schizophrenia With Duration of Illness < 10 Years
Brief Title: Paliperidone Extended Release in Schizophrenia Participants With Duration of Illness Less Than 10 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017578; R076477SCH3037; 2008-002384-13
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Results first posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone ER (Experimental)
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — Participants will be administered paliperidone extended release (ER) tablets orally (taken by mouth; to be swallowed) once daily in the dose range of 3 to 12 milligram (mg) for 13 weeks. Dose will be increased or decreased as per Investigator's discretion.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of paliperidone extended release (ER) in symptomatic participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) who were receiving treatment with any oral (having to do with the mouth) antipsychotic medication and who needed to be switched to paliperidone ER from the current oral antipsychotic therapy due to insufficient efficacy or due to side effects.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-centric (conducted in more than one center) and non-comparative study of paliperidone ER in participants with schizophrenia who have a previous history of bad adherence to the antipsychotic treatment because of insufficient efficacy and side-effects. All the eligible participants will receive a dose of paliperidone ER in range of 3 to 12 milligram (mg) orally (taken by mouth; to be swallowed) once daily for 13 weeks. Efficacy and safety will primarily be evaluated by Positive and Negative Syndromes Scale (PANSS) and Extrapyramidal Symptom Rating Scale (ESRS), respectively. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants meet the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria for schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self)
* Positive and Negative Syndrome Scale (PANSS) total score at Baseline of greater than equal to 70 and less than equal to 100
* Participants who need to be switched from the current oral antipsychotic therapy because of lack of efficacy or side effects
* Participants followed as outpatients
* Female participants must be postmenopausal for at least 1 year, surgically sterile or, if sexually active, be practicing an effective method of birth control and female participants of childbearing potential must also have a negative urine pregnancy test at Baseline

Exclusion Criteria:

* Acute psychotic relapse that requires hospitalization and first antipsychotic treatment ever
* Participants who had received clozapine during the previous 3 months
* History or current symptoms of tardive dyskinesia (twitching or jerking movements that you cannot control in your face, tongue, or other parts of your body) and neuroleptic malignant syndrome (high fever, rigid muscles, shaking, confusion, sweating more than usual, increased heart rate or blood pressure, or muscle pain or weakness)
* Pregnant or breast-feeding female
* Participated in an investigational drug trial in the previous 30 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A. Italy Clinical Trial, Study Director — Janssen-Cilag S.p.A.

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone ER: Participants were administered paliperidone extended release (ER) tablets orally (taken by mouth; to be swallowed) once daily in the dose range of 3 to 12 milligram (mg) for 13 weeks. Dose was increased or decreased as per Investigator's discretion.
Period: Overall Study
Arm/Group | Paliperidone ER
Started | 133
Completed | 118
Not Completed | 15
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 3
Not completed — Lost to Follow-up | 2
Not completed — Study medication non-compliant | 1
Not completed — Participant who withdrew consent | 8

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 132
Age Continuous [Mean (Standard Deviation); unit: years] — Out of a total of 133 participants, Baseline characteristic (Age) was available for only 132 participants who were included in intent to treat (ITT) population.
  years | 35.3 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants] — Out of a total of 133 participants, Baseline characteristic (Gender) was available for only 132 participants who were included in ITT population.
  Participants
    Female | 41
    Male | 91

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - Total Score at Week 13
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210, higher scores indicate worsening.
Time Frame: Baseline and Week 13
Population: Intent to Treat Population (ITT) included all participants who received at least 1 dose of study medication. For participants leaving study prematurely last available data post-baseline was used for final evaluation using Last observation carried forward (LOCF) method.' N' (number of participants analyzed): participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 126
units on a scale
  Baseline | 88.98 (10.126)
  Change at Week 13 | 22.468 (17.287)

2. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) - Positive Subscale Score at Week 13
Description: The PANSS Positive Subscale assesses seven positive-symptoms of schizophrenia. Positive symptoms refer to an excess or distortion of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology).
Time Frame: Baseline and Week 13
Population: The ITT included all participants who received at least one dose of study medication. For participants leaving study prematurely last available data post-baseline was used for final evaluation using LOCF method.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Paliperidone ER: Participants were administered paliperidone ER tablets orally (taken by mouth; to be swallowed) once daily in the dose range of 3 to 12 mg for 13 weeks. Dose was increased or decreased as per Investigator's discretion.
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 132
units on a scale
  Baseline | 21.03 (5.2)
  Change at Week 13 | -6.55 (5.3)

3. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - Negative Subscale Score at Week 13
Description: The PANSS Negative Subscale assesses seven negative-symptoms of schizophrenia. Negative symptoms represent a diminution or loss of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology).
Time Frame: Baseline and Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 132
units on a scale
  Baseline | 23.11 (6.4)
  Change at Week 13 | -4.82 (5.6)

4. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) General Psychopathology Subscale Score at Week 13
Description: The PANSS General Psychopathology Subscale Score assesses 16 general psychopathology symptoms. The symptoms are rated on a 7-point scale, with a range of 16 (absent) to 112 (extreme psychopathology).
Time Frame: Baseline and Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 132
units on a scale
  Baseline | 44.84 (6.5)
  Change at Week 13 | -11.31 (8.7)

5. Secondary Outcome: Percentage of Participants With Greater Than or Equal to 30 Percent Treatment Response in Total Positive and Negative Syndrome Scale (PANSS) Score
Description: as for outcome 1
Time Frame: Baseline and Week 13
Population: The ITT included all participants who received at least one dose of study medication. For participants leaving study prematurely last available data post-baseline was used for final evaluation using LOCF method. 'N' (number of participants analyzed) signified participants evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 126
percentage of participants | 40.5

6. Secondary Outcome: Change From Baseline in Subjective Well-being Under Neuroleptic (SWN 20) Scale at Week 13
Description: The SWN 20 scale is a 20 item scale that was originally designed to explore the subjective experience of psychotic participants. The SWN scale contains five sub-scales consisting of four items each: mental functioning (MF), self control (SC), emotional regulation (ER), and social integration (SI), physical functioning (PF). The total score ranges from a minimum of 20 (poor subjective experience) to a maximum of 120 (excellent subjective experience). SWN scores appear to correlate with measure of objective psychopathology, quality of life and other self-ratings of mood.
Time Frame: Baseline and Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 132
units on a scale
  Baseline | 73.81 (15.4)
  Change at Week 13 | 6.86 (12.8)

7. Secondary Outcome: Change From Baseline in Drug Attitude Inventory (DAI 30) Scale at Week 13
Description: The DAI is a 30-item self-rating inventory that focuses on subjective effects of neuroleptic medications in participants with schizophrenia. There are 15 items that are scored as true and 15 scored as false if the person is fully compliant (positive subjective response). Positive answers score as +1, negative answers score as - 1. Questionnaire allows identifying participants at high risk of low compliance. The total score may vary from -30 to +30 with a high total final score is a positive subjective response (compliant) and a low total score is a negative subjective response (non-compliant).
Time Frame: Baseline and Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 132
units on a scale
  Baseline | 41.20 (5.4)
  Change at Week 13 | 2.0 (5.4)

8. Secondary Outcome: Clinical Global Impression-Severity Scale (CGI-S)
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to normal, not at all ill and a rating of 7 is equivalent to among the most extremely ill participants. Higher scores indicate worsening.
Time Frame: Baseline and Week 13
Population: The ITT included all participants who received at least one dose of study medication. For participants leaving study prematurely last available data post Baseline was used for final evaluation using LOCF method.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 132
units on a scale
  Baseline | 4 [2 to 6]
  Week 13 | 3 [1 to 6]

9. Secondary Outcome: Change From Baseline in Personal and Social Performance Scale (PSP) at Week 13
Description: The PSP is 100-point validated clinician-rated scale that assesses degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors rated on 6-point scale (1=absent to 6=very severe).Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning, with higher transformed score indicating better function. Total score is divided into 3 levels: 71-100 (mild difficulty); 31-70 (marked difficulty) and 1-30 (severe difficulty).
Time Frame: Baseline and Week 13
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 132
units on a scale
  Baseline | 56.54 (12.47)
  Change at Week 13 | 9.05 (10.5)

10. Secondary Outcome: Quality of Sleep Score
Description: This self-administered scale rates quality of sleep and daytime drowsiness. Participants indicate on an 11-point scale how well they have slept in the previous 7 days, from 0 (very badly) to 10 (very well); and how often they have felt drowsy within the previous 7 days, from 0 (not at all) to 10 (all the time). On the sleep evaluation scale, score 0 corresponds to very badly and score 10 to very well.
Time Frame: Baseline and Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 132
units on a scale
  Baseline | 6.22 (2.5)
  Week 13 | 7.08 (2.1)

11. Secondary Outcome: Daytime Drowsiness Evaluation Scale
Description: This self-administered scale rates quality of sleep and daytime drowsiness. Participants will indicate on an 11-point scale how well they have slept in the previous 7 days, from 0 (very badly) to 10 (very well); and how often they have felt drowsy within the previous 7 days, from 0 (not at all) to 10 (all the time).On the daytime drowsiness scale, score 0 corresponds to not at all and score 10 to all the time.
Time Frame: Baseline and Week 13
Population: ITT included all participants who received at least one dose of study medication. For participants leaving study prematurely last available data post-baseline was used for final evaluation using LOCF method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 132
units on a scale
  Baseline | 4.09 (2.4)
  Week 13 | 3.30 (2.5)

12. Secondary Outcome: Extrapyramidal Symptoms Scale (ESRS) Subscale Scores and Total Scores
Description: Extra pyramidal symptoms attributed to antipsychotic assessed by ESRS scale. Included 4 subscales; Parkinsonism (Park),dystonia(Dyst),dyskinesia(Dysk),akathisia(Akat),12 items on 4-point scale; (0=absent-3=severe); Park (8 items); Dyst (2 items); Dysk (7 items) all 3 rated on 7-point scale (0=none/normal-6=worst). Additionally, subtotals were calculated; hyperkinesia (item 5, 6 of Park); hypokinesia (item 1-4, 7 of Park); bucco-linguo-masticatory (item 1-3 of Dysk), choreoathetoid movement (item 5, 6 of Dysk). Total score: sum of Park, Dyst & Dysk subscale, ranged from 0 (normal)-102 (severe).
Time Frame: Baseline and Week 13
Population: Safety population included all participants who received atleast one dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 132
units on a scale
  Baseline: ESRS Total Score | 7.39 (13.2)
  Week 13: ESRS Total Score | 2.21 (4.6)
  Baseline: Park, Dyst, Dysk and Akat | 1.86 (2.6)
  Week 13: Park, Dyst, Dysk and Akat | 0.56 (1.1)
  Baseline: Park | 4.30 (7.3)
  Week 13: Park | 1.33 (2.8)
  Baseline: Dyst | 0.66 (3.4)
  Week 13: Dyst | 0.15 (1.0)
  Baseline: Dysk Movements | 0.58 (1.7)
  Week 13: Dysk Movements | 0.18 (0.5)
  Baseline: Hyperkinesia | 1.43 (3.4)
  Week 13: Hyperkinesia | 0.44 (1.3)
  Baseline: Hypokinesia | 2.66 (4.4)
  Week 13: Hypokinesia | 0.80 (1.6)
  Baseline: Bucco-Linguo-Masticatory | 0.21 (0.7)
  Week 13: Bucco-Linguo-Masticatory | 0.05 (0.25)
  Baseline: Choreoathetoid movements of limbs | 0.20 (0.6)
  Week 13: Choreoathetoid movements of limbs | 0.06 (0.3)

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (Week 13)
Description: Safety population included all participants who receive at least one dose of study medication (n=132).
Arm/Group | Paliperidone ER
Serious Adverse Events (participants affected / at risk) | 1/132
Other Adverse Events (participants affected / at risk) | 21/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER (N=132)
Worsening of Schizophrenia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER (N=132)
Hypopiesia (Cardiac disorders) | 1
Increased Blood Pressure (Cardiac disorders) | 1
Tachicardia (Cardiac disorders) | 1
Rash (Mycosis) (Skin and subcutaneous tissue disorders) | 1
Galactorrhoea (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Weight Increase (Metabolism and nutrition disorders) | 4
Agitation (Nervous system disorders) | 1
Insomnia (Nervous system disorders) | 4
Akatisia (Nervous system disorders) | 1
Anxiety (Nervous system disorders) | 1
Extrapyramidal Symptoms (Nervous system disorders) | 3
Increased Anxiety (Nervous system disorders) | 1
Increased Irritability (Nervous system disorders) | 1
Jaw Movements (Nervous system disorders) | 1
Lingual Movements (Nervous system disorders) | 1
Lower Limbs Tremor (Nervous system disorders) | 1
Psychomotor Agitation (Nervous system disorders) | 1
Ptyalism (Nervous system disorders) | 1
Slowness (Increased) (Nervous system disorders) | 1
Worsening of Anxiety (Nervous system disorders) | 1
Worsening of Bradikinesia (Nervous system disorders) | 1
Worsening of Tremor (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days